CLINICAL TRIAL: NCT01315834
Title: The Contribution of Personality Traits to Marital Satisfaction, Well Being and Physical Health in Couples Coping With Coronary Heart Disease Versus a Control Group
Brief Title: Couples Coping With Coronary Heart Disease
Acronym: psychocardio
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10psycho-cardioCTIL
Record Dates: First submitted 2011-01-11; First posted 2011-03-15 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Heart Disease (CHD)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Couples coping with CHD: The target group will be 127 male patients and their partners. The couples will be recruited during the patients' first hospitalization for ACS. The participants will complete questionnaires during the hospitalization and again six months later. The patients will also be asked to be weighed and have their blood drawn and at the six-month follow-up for measurement of blood Cholesterol level. Relevant data will be obtained from their medical files.
- control group: The control group will be 100 couples who are not coping with a life threatening illness. The couples will complete self report questionnaires at one point of time.

SUMMARY:
The main purpose of this study is to examine the contribution of personality traits to marital satisfaction and well -being among couples coping with Coronary Heart Disease (CHD) and couples from the general population, and to health promoting behaviors and physical recovery among the ill partners.

DETAILED DESCRIPTION:
Heart disease is the world's leading cause of death in most industrial countries and it requires drastic changes in the lifestyle of the patient. Research on social support and coping with stress has repeatedly shown that being in a supportive spousal relationship has a significant effect on the recovery from a heart disease through alterations in mood, as well as through health habits. However, there are interpersonal differences in the abilities to receive and to provide support. Most of the literature to date has focused either on the experiences of the support recipient or on the support provider; much less research has taken both partners' characteristics into consideration (Revenson & DeLongis, 2011).

The current research aims to broaden the understanding of spousal support among couples coping with a life threatening illness- Coronary Heart Disease (CHD) versus general population of couples. Two studies were designed. Study 1(control group) will focus on general population of couples and its goal is examine the contribution of personality traits of the couples to their marital satisfaction and well-being. Study 2 (target group) will focus on couples coping with a first acute coronary heart disease and its goal is to examine the contribution of personality traits of the couples to their marital satisfaction and well-being, and to health promoting behaviors (smoking cessation, medication adherence) and physical recovery (change in body mass index, change in cholesterol levels) of the ill partners.

The proposed research is a prospective, longitudinal study. The control group will be 100 couples who are not coping with a life threatening illness. The couples will complete self report questionnaires. The target group will be 127 male patients and their partners. The couples will be recruited during the patients' first hospitalization for ACS. The participants will complete questionnaires during the hospitalization and again six months later. Relevant data will be obtained from their medical files.

This study's findings could inform clinicians whose goal is to foster better patient-spouse dynamics in the context of major medical stressors. Helping couples master the challenge of providing and receiving support in such trying times may contribute to enhanced levels of adherence among patients which, in turn, would lead to improved health and saved lives.

ELIGIBILITY:
Inclusion Criteria:

* Jewish men with a Clinical diagnosis of first Acute Coronary Syndrome (ACS: myocardial infarction (MI) or unstable angina (UA))
* Partners also agree to participate in the study

Exclusion Criteria:

* a history of a previous cardiac event
* a diagnosis other than ACS
* co-morbid conditions (such as a severe psychiatric illness, end state renal disease or severe cancer)
* absence of a spouse
* inability to be interviewed in Hebrew

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Paitents hospitalized Meir Medical Center Cardiac Care Unite
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Patients' medication adherence | Six months after hospitalization
  Medication adherence: the number of prescriptions filled as a function of the frequency of the medication. will be obtained from the central database of the patients' HMO.
Change in blood level Cholesterol | six mounths
  Change in blood level Cholesterol:Patients' blood level Cholesterol will be taken at baseline from their medical files and at the follow-up patients will be invited again for blood tests.
Change in body mass index | six-month
  Change in body mass index:Patients' BMI will be measured at baseline and Patients will be asked to weigh in again at the six-month follow-up
Smoking cessation | six months
  Smoking cessation:self-report measures of the patients'smoking cessation at follow-up.
Change in blood level Cholesterol | six mounths
  Change in blood level Cholesterol:Patients' blood level Cholesterol will be taken at baseline and at the follow-up from their medical files.

SECONDARY OUTCOMES:
Patients' and spouses' depression and anxiety symptoms | Case group- the instruments will be administered twice: at baseline and at the six- month follow-up Control group- the instruments will be administered at a one point of time
  Depression and anxiety- depressive and anxiety symptoms will be measured using the Brief Symptom Inventory [BSI;( Derogatis & Melisaratos, 1983)]. Each participant will be asked to rate the degree to which he has suffered from each symptom during the previous month on a scale ranging from 0 (not at all) to 4 (very much).
Patients' and spouses' marital satisfaction | Case group- the instruments will be administered twice: at baseline and at the six- month follow-up Control group- the instruments will be administered at a one point of time
  Marital satisfaction - marital satisfaction will be measured using the EMS-ENRICH Marital Satisfaction Scale (Lavee, 1995(.

CONTACTS AND LOCATIONS:
Overall Officials: Morris Mosseri, Professor, Principal Investigator — Department of Cardiology, Meir Medical Center, Israel
Locations (1):
- Department of Cardiology, Meir Medical Center, Kfar Saba, Israel